CLINICAL TRIAL: NCT04340388
Title: Contribution of the Integrase Inhibitor Dolutegravir to Obesity and Cardiovascular Disease in Persons Living With HIV
Brief Title: Contribution of Dolutegravir to Obesity and Cardiovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Jonell Poe, Assistant Clinical Professor, Physician Assistant, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1553691-1
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: HIV-1-infection; Antiviral Drug Adverse Reaction; Vascular Diseases; Cardiovascular Abnormalities; Abnormality of Adipose Tissue; Body Weight Changes; Body Fat Disorder; HIV-Associated Lipodystrophy Syndrome
MeSH Terms: conditions — Vascular Diseases; Cardiovascular Abnormalities; Body Weight Changes; HIV-Associated Lipodystrophy Syndrome | interventions — dolutegravir; tenofovir alafenamide; Tenofovir; abacavir; Lamivudine; Darunavir; Cobicistat; Rilpivirine; lamivudine, zidovudine drug combination; Zidovudine

STUDY DESIGN:
Intervention Model Description: The study design is a randomized control trial where patients will be randomized to the dolutegravir or non-dolutegravir arms by random number generation using the statistical software R. A unique identification (ID) key from 1 to 2n will be assigned to each patient.
  Additionally, the investigators will utilize a parallel mouse model of HIV mimicking PLWH with stable viral load that can provide mechanistic insight and integrate experiments at the tissue level (adipose tissue) as well. Experiments in the parallel mouse model of HIV will also present the advantage to enable the study the direct effects of HIV viral infection on metabolic and cardiovascular function, a study not feasible in PWH who, for easily understandable ethical reasons, cannot remain without treatment for 6 months (duration of the study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Switch from a non-integrase based regimen to dolutegravir (Active Comparator): Participants with HIV-1 infection who have had viral suppression on a non-integrase based antiretroviral regimen for greater than or equal to 3 months will be switched to a dolutegravir based regimen dosed at 50 milligrams (MG) once daily. Background regimen will remain the same.
  Interventions: Drug: Dolutegravir 50 MG
- Continue on non-integrase inhibitor based regimen (Active Comparator): Participants not currently on an integrase based regimen who remain on current suppressive therapy will remain on current antiretroviral regimen.
  Interventions: Drug: Antiretroviral/Anti HIV

INTERVENTIONS:
Drug: Dolutegravir 50 MG — 15 participants will be randomized to remain on fully suppressive background antiretroviral therapy. The third agent will be switched to dolutegravir at the dose of 50 mg daily.
  Other Names: Tenofovir alafenamide; Tenofovir disoproxil fumarate; Abacavir; Lamivudine; Darunavir; Cobicistat; Rilpivirine; Combivir; Zidovudine
  Arms: Switch from a non-integrase based regimen to dolutegravir
Drug: Antiretroviral/Anti HIV — 15 participants with suppressed HIV disease for greater than or equal to 3 months will be randomized to remain on their current 2 or 3 drug fully suppressive antiretroviral regimen.
  Other Names: Antiretroviral Combinations
  Arms: Continue on non-integrase inhibitor based regimen

SUMMARY:
The goal of the study is to combine a collaborative and translational approach to evaluate the effect antiretroviral regimen switch to a dolutegravir containing regimen compared to continued treatment with a non- dolutegravir based regimen on on lipid and metabolic profiles, renal function, body composition, vascular function and diet.

DETAILED DESCRIPTION:
Over the last decades, the use of combined antiretroviral therapy has led to profound suppression of HIV-1 replication and increased the survival of persons living with HIV (PLWH) to close to that of the general population. As a consequence, the spectrum of diseases related to HIV has shifted from opportunistic AIDS-related diseases towards long-term-age-related complications. Individuals living with HIV are now exhibiting accelerated development of obesity, metabolic derangements and cardiovascular disease (CVD). Recent compelling clinical evidence has documented a drastic shift in anthropometric profiles among persons living with HIV. In addition, several reports present dolutegravir, a second-generation integrase inhibitor currently highly prescribed for its high antiviral efficiency, as the potential cause of unpredicted weight gain. A critical gap in the investigators' knowledge is a lack of understanding of the etiopathology of the contribution of dolutegravir on weight gain and the consequential impact on obesity and cardiovascular disease in persons living with HIV on combined antiretroviral therapy. As overweight and obesity are among the leading risk factors for cardiovascular disease in persons living with HIV, it is critical to directly investigate whether dolutegravir increases fat mass in persons living with HIV and whether body weight gains-associated with dolutegravir based regimen contribute to the increased prevalence of CVD in this population of people.

This application seeks to investigate alterations in body fat and cardiometabolic risk markers associated with dolutegravir. The investigators propose that in patients with undetectable plasma HIV RNA, there is a direct correlation of weight gain and dolutegravir after antiretroviral regimen switch. They also contend that dolutegravir associated weight gain induces a phenotypic metabolic shift which alters the vascular endothelium and potentiates CVD risk. If the investigators are correct in their hypotheses, modifications in the clinical practice of treatment and prevention strategies for CVD in people living with HIV may be warranted.

Herein the investigators propose a novel translational study which will concomitantly investigate in human patients and animal models of HIV:

1. whether dolutegravir based regimen increases body weight
2. the mechanisms whereby dolutegravir increases body weight
3. whether dolutegravir-mediated body weight gain increases the risk for CVD in PLWH.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for participation in this study:

* Age greater than or equal to 18 years with HIV-1 who have been virologically suppressed (HIV-1 RNA < 50 copies for greater than or equal to 3 months on a non-integrase strand transfer inhibitor-based regimen
* Have the ability to understand and sign an informed consent written in the English language

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in this study:

* Age less than 18 years without HIV-1 infection
* Has hypersensitivity or other contraindication to any of the components of the study
* Has active diagnosis of untreated hepatitis due to any cause
* Has a history or current evidence of any condition, laboratory abnormality or other circumstance ( including drug or alcohol use or dependence) that might confound the results of the study or interfere with the subject's participation for the full duration of the study
* Is taking or is anticipated to require long term systemic immunosuppressive therapy, immune modulators, or any prohibited therapies from 60 days prior to Screening/Day 1 visit through to the end of study
* Has documented or suspected dolutegravir-associated resistance mutations specifically:

Q148H/K/R/N in combination with E138K or G1402/A or N155H.

* Has a life expectancy less than or equal to one year
* Is pregnant, breastfeeding, or expecting to donate eggs or sperm or conceive or father a child at any time during the study and 6 weeks following the end of study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 24 weeks
  Change from baseline kilograms (kg) of weight at 24 weeks

SECONDARY OUTCOMES:
Change in body mass index (BMI) | 24 weeks
  Total change in body mass index -height and weight will be combined to report BMI (Kilogram/Height in centimeters^2)
Change in vascular endothelial function | 24 weeks
  Change from baseline vessel diameter (millimeters) at 24 weeks
Height | 24 weeks
  Measurement of height (centimeters) from baseline to 24 weeks

OTHER OUTCOMES:
Change in cholesterol | 24 weeks
  Change from baseline cholesterol (mg/dL) at 24 weeks
Change in triglycerides | 24 weeks
  Change from baseline triglycerides (mg/dL) at 24 weeks
Change in high density lipoprotein (HDL) | 24 weeks
  Change from baseline HDL (mg/dL) at 24 weeks
Change in low density lipoprotein (LDL) | 24 weeks
  Change from baseline LDL (mg/dL) at 24 weeks
Change in HIV-1 RNA viral load | 24 weeks
  Change from baseline HIV-1 viral load (copies) at 24 weeks
Change in fasting serum glucose level | 24 weeks
  Change from baseline serum glucose level (mg/dL) at 24 weeks
Change in quantity of food consumption | 24 weeks
  Change from baseline of calorie consumption (kcal) at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonell B Poe, MPAS, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified all IPD included in this study and that de-identified IPD results that underlie applications for additional funding or for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following publication. No end date.
Access Criteria: To achieve aims in the approved proposal.

REFERENCES:
- [Result] Cottrell ML, Hadzic T, Kashuba AD. Clinical pharmacokinetic, pharmacodynamic and drug-interaction profile of the integrase inhibitor dolutegravir. Clin Pharmacokinet. 2013 Nov;52(11):981-94. doi: 10.1007/s40262-013-0093-2. PMID 23824675